CLINICAL TRIAL: NCT06867146
Title: The Role of Molecular Residual Disease in the Treatment Strategy and Prognosis Prediction of Pancreatic Cancer Patients Undergoing Adjuvant Therapy
Brief Title: MRD in PAAD Adjuvant Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K3378
Record Dates: First submitted 2024-11-18; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: The Role of Molecular Residual Disease in the Treatment Strategy and Prognosis Prediction of Pancreatic Cancer Patients Undergoing Adjuvant Therapy; Molecular Residual Disease; Pancreatic Cancer; Adjuvant Therapy
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: For patients with pathological stage I pancreatic cancer, if they are baseline MRD-positive after surgery, or MRD-negative but have high-risk recurrence factors (including perineural invasion, lymphovascular invasion, preoperative CA19-9 > 180 U/ml, postoperative CA19-9 > 37 U/ml, or extrapancreatic tumor infiltration), they will receive standard dual-agent chemotherapy, such as gemcitabine combined with nab-paclitaxel or capecitabine, with the chemotherapy regimen selected by the clinical doctor. If the patient is baseline MRD-negative and has no high-risk recurrence factors, they will be randomly assigned in a 1:1 ratio to either receive standard chemotherapy or be observed.
  For patients with pathological stage II-III pancreatic cancer, if they are baseline MRD-negative after surgery, they will receive standard dual-agent chemotherapy, such as gemcitabine combined with nab-paclitaxel or capecitabine, with the chemotherapy regimen selected by the clinical doctor. If the patient is ba
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD postive (Sham Comparator)
  Interventions: Drug: Three-drug chemotherapy group
- MRD negative (Active Comparator)
  Interventions: Drug: two-drug chemotherapy group

INTERVENTIONS:
Drug: Three-drug chemotherapy group — Three-drug chemotherapy group, mFOLFIRINOX, including 5-fluorouracil, leucovorin, oxaliplatin and irinotecan.
  Arms: MRD postive
Drug: two-drug chemotherapy group — two-drug chemotherapy group, including gemcitabine-based combination regimens (predominately gemcitabine/nab-paclitaxel or gemcitabine/capecitabine)
  Arms: MRD negative

SUMMARY:
Our preliminary research has explored the detection efficacy of minimal residual disease (MRD) in pancreatic cancer. In patients with pancreatic cancer undergoing dual-agent adjuvant chemotherapy, the median recurrence-free survival (RFS) is approximately 13.9 months. Due to the high postoperative recurrence rate, short survival time, and intense systemic chemotherapy in pancreatic cancer patients, there is an urgent clinical need to more accurately identify which patients will benefit from adjuvant therapy. This study aims to evaluate the application value and guiding significance of peripheral blood MRD in the decision-making process for adjuvant treatment in patients with resected pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Here's the translated and polished version of your content:

  1. Patients clinically diagnosed with pancreatic cancer, staged I-III (AJCC V8.0), who are scheduled to undergo curative surgery.
  2. No restrictions on gender; age between 18 and 70 years.
  3. Eastern Cooperative Oncology Group (ECOG) performance status score: ≤2.
  4. Expected survival time of ≥3 months.
  5. Willingness to comply with the study protocol for testing, treatment, and follow-up; consent to provide necessary clinical, pathological, and follow-up data for the study; and agreement to use the research data for future studies and product development.
  6. Voluntary participation in this clinical study, with an understanding of the study procedures and the ability to sign an informed consent form.

Exclusion Criteria:

1. Patients who have had other malignancies within the five years prior to this study.
2. Patients who have received any antitumor treatment within six months prior to enrollment.
3. Patients with concomitant diseases that, in the investigator's judgment, pose a serious risk to patient safety or could affect the patient's ability to complete the study (such as poorly controlled hypertension, severe diabetes, thyroid disorders, psychiatric disorders, etc.), or any other conditions deemed unsuitable for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
DFS | up to 18 months
  DFS refers to the length of time after treatment during which a patient remains free of any signs or symptoms of the disease. It is primarily used in cancer research to measure the effectiveness of treatments in preventing recurrence. Median follow-up time up to 18 months

SECONDARY OUTCOMES:
OS | up to 18 months
  OS measures the length of time from either the diagnosis or the start of treatment to the death of the patient, regardless of cause. Median follow-up time up to 18 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China